CLINICAL TRIAL: NCT07213661
Title: Long-term Comparative Effectiveness of 2 Treatments to Arrest Dental Caries in Older Adults
Brief Title: LT Comparative Effectiveness of 2 Caries Treatments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Suchitra Nelson, Associate Dean of Clinical and Translational Research Professor and Interim Chair, Community Dentistry, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20250955; LTF-2024C2-39677 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-10-03; First posted 2025-10-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries
Keywords: Dental Caries; Oral Health Quality of Life; Tooth Loss
MeSH Terms: conditions — Dental Caries; Tooth Loss | interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Intervention Model Description: The interventions will be continued in this long-term follow-up study for any new decay. Both coronal and root surface tooth decay lesions will be treated. The two evidence-based strategies in older adults will be compared as follows:
  Intervention Arm 1: A "simple medical strategy" consisting of SDF Participants will receive bi-annual application of topical 38% silver diamine fluoride (Advantage Arrest, Elevate Oral Care LLC., West Palm Beach, FL) following manufacturer's instructions and guidelines published by UCSF.
  Control Arm 2: A "typical dental strategy" consisting of ART + FV Atraumatic Restorative Treatment (ART) will be a modification of the approach used by Lo and colleagues (2006),2 and the cavity restored at baseline with resin reinforced glass-ionomer cement (GIC) (GC Corporation, Japan).
  Participants in this arm will also receive biannual topical fluoride varnish application (FluoriMax, Elevate) according to manufacturer's instructions.
Who Masked: Participant
Masking Description: We will maintain blinding of participants to the study arm but this may not be possible due to SDF color change. Clinical and study staff cannot be blinded due to the nature of the interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- A "simple medical strategy" consisting of SDF (Experimental): This treatment will be a bi-annual application of 38% silver diamine (Advantage Arrest, Elevate Oral Care LLC., West Palm Beach, FL) solution to new ICDAS lesions code 3-6 (at baseline and 26-weeks or 26-weeks and 52 weeks) following manufacturers instructions and guidelines published by UCSF (2016).
  Interventions: Device: A "simple medical strategy" consisting of silver diamine fluoride (SDF)
- A "typical dental strategy" consisting of ART + FV (Active Comparator): Atraumatic Restorative Treatment (ART) will be a modification of the approach used by Lo and colleagues (2006),2 and the cavity restored at baseline with resin reinforced glass-ionomer cement (GIC) (GC Corporation, Japan).
  Participants in this arm will also receive biannual topical fluoride varnish application (FluoriMax, Elevate) according to manufacturer's instructions.
  Interventions: Device: A "typical dental strategy" consisting of atraumatic restorative treatment (ART) with glass ionomer cement + Fluoride Varnish (FV)

INTERVENTIONS:
Device: A "simple medical strategy" consisting of silver diamine fluoride (SDF) — Bi-annual topical application of 38% silver diamine solution to new ICDAS lesions code 3-6. Advantage Arrest, Elevate Oral Care, West Palm Beach FL
  Other Names: SDF Treatment
  Arms: A "simple medical strategy" consisting of SDF
Device: A "typical dental strategy" consisting of atraumatic restorative treatment (ART) with glass ionomer cement + Fluoride Varnish (FV) — GC Fuji (for ART) and FluoriMax Varnish. Atraumatic Restoration Treatment (ART) to new ICDAS lesions code 3-6, followed by bi-annual topical fluoride varnish (FV) to all teeth.
  Other Names: ART + FV Treatment
  Arms: A "typical dental strategy" consisting of ART + FV

SUMMARY:
This study is a continuation of a cluster randomized clinical trial (cRCT) conducted in 33 publicly subsidized housing facilities/sites (HUD Section 202) and other low-income housing voucher programs in NE Ohio. The Intervention Arm (18 sites) - participants received biannual silver diamine fluoride (SDF) versus the Control Arm (15 sites) where participants received atraumatic restorative treatment (ART) with glass ionomer cement (GIC) + biannual fluoride varnish (FV) application. A total of 568 participants were recruited in the original study, and 480 participants (Intervention Arm: 287, Control Arm: 193) are expected to continue in this long-term follow-up study. Since enrollment in the original study was done over time, each participant will contribute data at 3 to 6 years (from randomization) in the LTFU depending on study entry to assess clinical equipoise of the two treatments.

Community-dwelling older adults, regardless of medical, cognitive, or motor impairments, were considered for inclusion in the original study and were: (1) aged ≥ 62 years in the 33 housing facilities; (2) have at least one untreated active root or coronal carious lesion with ICDAS-II lesion severity code of 3 or greater ; (3) willingness to stay in the study for 1 year. Exclusion criteria: (1) sensitivity to silver or other heavy-metal ions; (2) serious life-threatening medical disease. Additionally, any participant with the presence of gingival/perioral ulceration or stomatitis or tooth abscess in any specific tooth were referred to a dentist and enrolled after resolution. The LTFU study will follow the same enrolled participants long-term. The current mean (sd) age of the 480 participants who will enter the LTFU study will be 73.73 (6.92) years.

DETAILED DESCRIPTION:
Study Design: The original design was a cluster randomized clinical trial (RCT) in 33 publicly subsidized housing facilities/sites in NE Ohio and housing sites randomized into 2 arms in a roughly 1:1 ratio (SDF vs. ART + FV) and is a continuation of the original study "Reducing Oral Health Disparities of Older Adults: Comparative Effectiveness of 2 Treatments". All participants will be followed for one year and will receive intervention when new decay is present. The study hypothesis for the LTFU study is noninferiority of SDF to ART + FV for each of the primary outcomes. Primary outcomes are assessed through clinical and questionnaire evaluations. We will maintain blinding of participants to the study arm. Other clinical and study staff cannot be blinded due to the nature of the interventions.

Study Population and Setting: For the Intervention Arm, a total of 287 participants from 18 facilities will receive biannual 38% SDF, and for the Control Arm, a total of 193 participants from 15 facilities will receive ART + biannual FV application for new decay. Housing sites are located in three counties in Northeast Ohio (Cuyahoga, Summit, and Lorain). IRB approval was given allowing study staff to contact participants from the original study for future studies. Informed consent for LTFU will be obtained in-person at scheduled "Dental Days" at the housing sites. These will be scheduled in coordination with the housing site Service Coordinators, who will be briefed well in advance of LTFU activities.

A total of 480 participants (out of 568 from the original study) are expected to be retained into the LTFU study. Among the 480 participants to be consented and enrolled in the long-term follow-up, 26% (n-124), 36% (n=173), 17% (n=82), 21% (101) will contribute data at 3, 4, 5, 6 years post-randomization respectively. Each participant will be followed for one year (total of 3 visits -baseline (LTFU #1), 26 weeks (LTFU #2), 52 weeks (LTFU #3).The study population are predominantly low socioeconomic status (SES) and are adults ≥ 62 years of age residing in 33 participating HUD Section 202 and other publicly subsidized housing facilities. The population is diverse: African American/Black, Caucasian/White including Hispanic/Latino, and Asian. Medicaid participation among the tenants is 76% among facilities. The characteristics of the 480 in this long-term follow-up vs. the 568 participants that completed the cRCT are similar as follows: mean age 69.5±6.6 vs. 69.6±6.8; female 52% vs. 51%; Hispanic 2.9% vs. 2.7%; black 66% vs. 66%, white 29.6% vs. 29.3%; high school education or less 57% vs. 57.2%; living alone 93.7% vs. 93.3%; annual income $12, 490 or less 53.4% vs. 53.1%. Bi-variate analysis of the 480 LTFU participants vs. 88 non-participants indicate no significant differences in any of the characteristics indicating representativeness of the LTFU study population. These participants are also a diverse representation of the overall population in NE Ohio.

Analytic Plan: Analyses will follow the intent-to-treat principle; namely, the SDF and ART groups to be compared will be defined according to the randomization of sites (and original site residency of individuals). Preliminary analyses will involve the construction of one-sided 95% confidence interval based on a t-test (or other appropriate test) for the difference in mean responses (ART minus SDF) at selected long-term follow-up times. To account for clustering, a modified approach for these t-tests to allow for a possible non-zero within-facility correlation will be used. If this confidence interval lies below (for an outcome where higher is better) or above (where lower is better) the tolerance value then we may make the preliminary conclusion of 'non-inferiority' of SDF relative to ART with respect to that outcome. Confidence intervals will also be used to determine superiority of one intervention relative to the other.

To corroborate initial results, we will conduct generalized estimating equations (GEE) analyses. Specifically, for each outcome at the targeted long-term follow-up time, we will fit a GEE (marginal) model including, as covariates, an indicator variable for treatment and a selected set of baseline variables (including sociodemographic - e.g., race, gender and age, medical conditions, and oral health behavior variables) that are prognostic for the given outcome. Appropriate link functions will be used: a logit link for binary or binomial outcomes (including the arrest rate), a log link for count outcomes (number of newly missing teeth and number of newly decayed teeth), and an identity link for continuous outcomes (tooth pain score and GOHRQoL). An exchangeable working correlation matrix will be used to account for correlations among subjects within site. Inferiority and superiority (based on appropriate - possibly scale-transformed - tolerance values) will be tested using robust t tests with correction for a small number of clusters (or via corresponding 95% confidence intervals).

Secondarily, we will apply, to the repeated measures of each outcome (including initial study as well as long-term follow-up measurements) extended GEE models that include (in addition to the above mentioned covariates) time and possibly a time by treatment interaction, as well as an appropriate within-site working correlation structure (e.g., including an autocorrelation structure for the repeated measures over time). For each outcome model, we will estimate and test, via a robust t-test, the time by intervention interaction term to compare trends of the mean outcome over time for the two interventions; we will also separately assess intervention effects at multiple times in the long-term follow-up as well as consider more complex trends, e.g., including a quadratic time term. The same approach as above will be conducted for the secondary outcome, gingival inflammation. In that case, being a continuous outcome, an identity link will be used in the GEE model.

Sensitivity Analyses: We will check sensitivity of conclusions to model assumptions as well as methodological decisions such as outcome definition. For the GEE analyses, sensitivity will be assessed in part by using alternative working covariance structures and (for repeated measures analyses) alternative functions of time. For some outcomes, alternative distributions will be considered; for example, for count outcomes such as number of newly missing teeth, we will consider Poisson, negative binomial, zero-inflated Poisson (ZIP), and zero-inflated negative binomial (ZINB) distributions. Sensitivity to assumptions regarding missing data will also be investigated as described further below.

Missing Data: (a) Methods to prevent and monitor missing data: All questionnaires (using tablets) and dental assessment forms (using paper), will be managed in an electronic database (REDCap) by study staff. Weekly quality control checks will be run for outliers, entry errors, missing data, and potential data anomalies. Statistical analyses, summary and missing data reports will be generated by the study biostatistician monthly during the study. (b) Statistical Methods to Handle Missing Data and Account for Statistical Uncertainty Due to Missingness: In the preliminary approach, we will utilize complete cases for included baseline variables and will use all available measurements of each outcome for each individual; this approach assumes missing completely at random (MCAR) data, that is, missingness related only to baseline variables. In additional, a multiple imputation approach will be conducted as described below. (d) Plans to Record and Report Dropout and Missing Data: The trial data will be managed using REDCap electronic data capture platform as in the original study. REDCap is a secure web-based application providing an intuitive interface for validated data entry, audit trails for tracking data manipulation and export procedures, and automated export procedures for seamless data downloads to common statistical packages. Missing data reports will be generated weekly from REDCap for timely resolution and reporting purposes. (e) Plans to Examine Sensitivity of Inferences to Missing Data Methods: The MCAR assumption seems reasonable for missingness due to variation in measurement times (which depend on when the subjects entered the initial study), but more questionable for missingness due to death or other causes of dropout. We will test for a relationship between missingness and available (earlier) outcomes to evaluate the plausibility of the MCAR assumption. As a sensitivity analysis, we will conduct multiple imputations (relaxing MCAR and making the missing at random, MAR, assumption), for example using the multiple imputation by chained equations (MICE) algorithm with an appropriate imputation model, e.g., using logistic regression or predictive mean matching) depending on the type of outcome.

Reporting Plan: To allow for assessment of study's internal and external validity, we will adhere to standard reporting guidelines for randomized clinical trials as specified by: EQUATOR network; SPIRIT 2013 statement; and CONSORT 2010 statement.

ELIGIBILITY:
Inclusion Criteria: To be eligible to participate in this study, an individual must meet all of the following criteria:

* Were participants in the original study from the 33 housing sites
* Provide signed and dated long-term follow-up informed consent form
* Willingness to stay in the LTFU study for 1 year
* Additionally for focus groups, completed the treatment phase of the study

Exclusion Criteria: An individual who meets any of the following criteria will be excluded from participation in this study:

* Sensitivity to silver or other heavy-metal ions
* Serious life-threatening medical disease
* Additionally, any participant with the presence of gingival/perioral ulceration or stomatitis or tooth abscess in any specific tooth will be referred to a dentist but can only be enrolled after resolution

Min Age: 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Caries Arrest Rate | Baseline (LTFU 1) to 52-weeks (LTFU 3)
  ICDAS examinations are used to assess caries arrest on permanent tooth surfaces with moderate to severe lesions (ICDAS codes 3-6 with activity code 2) that received SDF or ART + FV treatment. A lesion is considered arrested if, at follow-up, the activity code is 1 (inactive) or the surface is sound (code S). The overall mean will be calculated by surfaces.
New Decay Rate | Baseline (LTFU 1) to 52-weeks (LTFU 3)
  New decay is defined as ICDAS lesion code ≥3 (localized to extensive decay) on one or more surfaces on newly decayed teeth found at LFTU #1, #2 and #3 (even on surfaces that did not receive the study treatments). The overall mean of decayed surfaces will be calculated.
Tooth Loss | Baseline (LTFU 1) to 52-weeks (LTFU 3)
  Tooth loss will be assessed through ICDAS exams by documenting absence of teeth. The overall mean will be calculated for the number of teeth lost.
Tooth Pain | Baseline (LTFU 1) to 52-weeks (LTFU 3)
  Tooth Pain and Sensitivity will be assessed using the PROMIS v.1.0 - Pain Intensity 3a [Modified for Dental]. An overall mean pain intensity score will be created for the 3-item Likert scale with answers ranging from 0-no pain to 4-very severe.
Oral Health Related Quality of Life | Baseline (LTFU 1) to 52-weeks (LTFU 3)
  Geriatric Oral Health Related Quality of Life (GOHRQoL) is an overall score created by taking the sum of each of the 12 items, which are on a Likert scale using 3 levels (Always/Often - 1, Sometimes/Seldom - 2, Never - 3). The scores range from 12-36 with higher scores indicating better quality of life. The overall mean for the participant population will be calculated.

SECONDARY OUTCOMES:
Gingival Inflammation Index | Baseline (LTFU 1) to 52-weeks (LTFU 3)
  Gingival inflammation will be assessed using the Modified Gingival Index. Scores range from 0-4, with 0 being healthy gums, 1-mild inflammation, 2-moderate inflammation, and 3 and 4 (more bleeding and ulceration) being severe inflammation. The mean overall scores will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra S Nelson, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No